CLINICAL TRIAL: NCT01879995
Title: Nutrition Status of Adult and Adolescent Patients With Classical Phenylketonuria (PKU) and Hyperphenylalaninemia
Brief Title: Phenylketonuria and Hyperphenylalaninemia Nutrition Study
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2013-0120
Record Dates: First submitted 2013-06-04; First posted 2013-06-18 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Phenylketonuria (PKU) and Hyperphenylalaninemia
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Procedure:

SUMMARY:
The mainstay of PKU treatment is a low-phenylalanine diet (i.e restriction of natural protein), and supplementation with a protein substitute (a mixture of amino acids free from phenylalanine, also containing micronutrients and vitamins) and special low-protein foods, to meet the patient's energy requirements. When diet and treatment is relaxed after childhood, adult and adolescent patients with phenylketonuria are at risk for malnutrition, depending on the compliance with treatment and the intake of amino acid supplements.

In this study, nutrition status of patients with PKU and hyperphenylalaninemia is systematically assessed under ongoing current treatment, in relation to Phe-tolerance, compliance with treatment, and psychosocial issues.

Study participants do not undergo any specific therapeutic or diagnostic intervention.

ELIGIBILITY:
Inclusion criteria:

* PKU (Phenylketonuria) or hyperphenylalaninemia
* male or female, minimum age 16y
* signed informed consent

Exclusion criteria:

- patient who can not comply with the study protocol (e.g. unable to fill in questionnaires by themselves or a representative)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with phenylketonuria or hyperphenylalaninemia, in treatment at the participating centres
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Macronutrient and micronutrient intake, calculated from a nutrition protocol (four consecutive days) | assessed during 4 consecutive days max. within 1 month after a regular consultation in the outpatient clinic
  Assessed nutrients:
  Macronutrients: protein, fat, carbohydrates in g/kg/d
  Daily phenylalanine and tyrosine intake Micronutrients and minerals: Calcium, magnesium, iron, zinc, selenium
  Vitamins: D, B12, B6, C, folic acid

SECONDARY OUTCOMES:
Phenylalanine level (umol/l) | assessed at the end of the four-day nutrition protocol (see primary outcome)
  this outcome measure is not study-specific and is collected as part of established routine care (self-measurement by patient)
Plasma amino acid profile | determined at a routine visit at the outpatient clinic, on average 1x per year
  this outcome measure is not study-specific and is collected as part of established routine care.
Concentrations of micronutrients, minerals and vitamins | determined at a routine visit at the outpatient clinic, on average 1x per year
  assessed parameters: Ferritin, zinc, selenium, vitamin D, vitamin B12, folic acid.
  These outcome measures are not study-specific and are collected as part of established routine care
body weight (kg) | determined at a routine visit at the outpatient clinic, on average once every 6 - 12 months
  assessed as part of routine clinical care

CONTACTS AND LOCATIONS:
Overall Officials: Michel Hochuli, MD PhD, Principal Investigator — University Hospital Zurich, Division of Endocrinology, Diabetes and Clinical Nutrition
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Division of Endocrinology, Diabetes and Clinical Nutrition, Zurich, Canton of Zurich
  - University Children's Hospital, Zurich